CLINICAL TRIAL: NCT06637618
Title: Cluster and Registry Trial Of the Working Group of Heart Failure in Denmark. Does the Strategy of Initiation of Heart Failure Medication Matter in the Real World.
Brief Title: Does the Sequence of Heart Failure Medication Matter
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Hillerod Hospital, Denmark (Other); Herlev and Gentofte Hospital (Other); Slagelse Hospital (Other); Bispebjerg Hospital (Other); Naestved Hospital (Other); Svendborg Hospital (Other); Sygehus Lillebaelt (Other); Aabenraa Hospital (Other); Viborg Regional Hospital (Other); Randers Regional Hospital (Other); Regionshospitalet Silkeborg (Other); Regionshospital Nordjylland (Other Government); Hospitalsenheden Vest (Other)
Responsible Party: Principal Investigator, Mads Jønsson Andersen, Senior Registrar, MD PhD, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CROWD sequence
Record Dates: First submitted 2024-09-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Heart Failure, Reduced Ejection Fraction
Keywords: heart failure; pharmacology; cluster randomised controlled clinical trial; mineralocorticoid receptor antagonist; beta blocker; ace inhibitor; sglt2 inhibitor
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure

STUDY DESIGN:
Intervention Model Description: An open-label cluster randomised crossover clinical trial, assessing the effect of upfront use of mineralocorticoid antagonists versus usual sequencing of heart failure medication
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard care (Active Comparator): standard care, with physicians choice of the sequence and up-titration of heart failure medications (ACE-inhibitor, beta-blocker, mineralocorticoid receptor antagonist, SGLT2-inhibitor)
  Interventions: Behavioral: up front use of mineralocorticoid receptor antagonist
- Up-front prescription of mineralocorticoid receptor antagonist, no later than the first ambulatory v (Experimental): Up-front prescription of mineralocorticoid receptor antagonist, no later than the first ambulatory visit to the heart failure clinic. Earlier use during initial hospitalization is encouraged, but not mandatory
  Interventions: Behavioral: up front use of mineralocorticoid receptor antagonist

INTERVENTIONS:
Behavioral: up front use of mineralocorticoid receptor antagonist — the sequence of which the four drug classes are prescribed will differ, where the intervention is early use of MRA, where the control group will receive standard care, where MRA are usually prescribed last

SUMMARY:
This study will tests whether a strategy of upfront prescription of mineralocorticoid receptor antagonists (MRA) is different from usual care, where MRA are usually prescribes as the last drug of the four drug classes used in the treatment of heart failure with reduced cardiac pump function (ace-inhibitor, beta blocker, sodium-glucose-2 inhibitors, MRA).

The study is a national study that intends to include all adult Danish patients diagnosed with heart failure and reduced pump function from early 2025 til early 2029.

Treatment strategy will be decided by randomisation, where each heart failure clinic is randomised to one of the two strategies (upfront MRA vs. usual care) for one year, followed by cross-over to the other treatment strategy for one year.

Patients will be followed according to usual care at their respective heart failure clinic. Study-specific followup will be conducted through the Danish registries for a minimum of two years.

The primary goal of the study is to evaluate whether one of the two treatment strategies leads to fewer hospitalisations for heart failure and/or death at one year after study entry.

Other goals of the study is to evaluate whether one of the two strategies leads to less kidney disease, improved quality of life and improved cost-effectiveness

DETAILED DESCRIPTION:
This study aims to examine whether upfront initiation of MRA followed by usual care of HFrEF medication up-titration with ACE or ARB, SGLT2 inhibitors, and beta-blockers can improve clinical outcomes compared to the usual care approach (ACEi/ARB or ARNi, BB, SGLT2i followed by MRA). The investigators hypothesize that upfront initiation of MRA may enhance adherence to MRA therapy. To test this hypothesis, a cluster randomized controlled trial will be performed comparing two strategies: [1] upfront initiation of MRA followed by usual care of up-titration of HFrEF medication versus usual car (ACEi/ARB or ARNi, BB, SGLT2i followed by MRA). This study will provide valuable insights into whether upfront initiation of MRA impacts patient outcomes, potentially leading to a shift in HFrEF management.

Methods

Design CROWD-Sequence is a cluster-randomized crossover comparative effectiveness study.

Intervention All patients will receive treatment according to national guidelines, which include all 4 pillars of modern HFrEF treatment. The intervention is only whether the heart failure clinic initiates MRA upfront at the first visit, compared with the initiation of MRA later in the up-titration of HFrEF medication.

Cluster allocation Each participating heart failure clinic will be allocated to four periods (clusters): two periods with upfront initiation of MRA followed by usual care of HFrEF medication and two periods with usual care of up-titration of HFrEF medication with initiation of MRA at a later stage. Heart failure clinics will be randomly allocated and alternate between the two strategies annually. The estimated total participation time for each heart failure clinic is four years. The randomization is unblinded. Randomization of the heart failure clinics will be performed in a 1:1 fashion. Details of randomization and allocation periods will be stored at the Sponsor.

If a cluster is scheduled to stop before two years due to organizational changes (e.g., if the heart failure clinic is closed or merged with another clinic), the investigators may change the duration of the remaining periods for that cluster to get compatible allocation periods.

Eligible departments Danish cardiology departments with a heart failure clinic reporting to the Danish Heart Failure Registry are eligible. All responsible contact persons are listed in Appendix 1. Each contact person will comply with the protocol-requirements. Further, all 26 heart failure clinics will have the same inclusion and exclusion criteria regardless of their cluster allocation.

Eligible patients

Patients will be identified when registered in the Danish Heart Failure Registry. All patients ≥18 years old who are newly diagnosed with HFrEF and are allocated to an outpatient clinic for up-titration of guideline-directed medical therapy for HFrEF at participating cardiology departments are candidates for the study. Patients will be informed about the study and given the option to opt out of all analyses.

The criteria for being included in the Danish Heart Failure Registry are described in Schjoedt et al., 2016. [11] In brief, patients enrolled in the registry must be 18 years or older and have a first-time hospital contact with heart failure as the primary diagnosis using the European Society of Cardiology criteria.

Information to the patients

Eligible patients will be informed about the trial through posters and flyers within the department. Their treating physician or nurse will inform them directly when initiating the HFrEF medication. They will be informed that the department is part of a national effort to compare two similar strategies and will be briefed on the specific strategy currently employed by the heart failure clinic. Patients will have the opportunity to opt out of all analyses. Those who choose to opt out will be registered in a nationally accessible REDCap database.

Treatment in allocation arms

Treatment in clusters will adhere to both Danish and European guidelines. The treating physicians will treat patients according to general clinical practice. The randomization is only regarding at what time point MRA is initiated, not the actual drug prescribed. The guideline-recommended treatment will adhere to both Danish and European guidelines. The treating physicians will treat patients according to general clinical practice. If a patient has a contraindication for a specific drug class (e.g. hypersensitivity to the active substance etc.), then the patient will not be prescribed this class of drugs. An instrumental variable analysis in the per-protocol analysis will be used to allow for this potential confounding by (contra)indication. There will not be any extra patient visits due to the study, and there will not be any increased economic burden on the patient.

Information to the departments about activities in the trial and treatment allocation

Heart failure clinics will be instructed in the activities of the trial in three ways: 1) all contact persons at each heart failure clinic will be sent the protocol together with written instructions on the conduct of the trial; 2) all heart failure clinics will be offered an individual meeting on the conduct of the trial; and 3) during the trial, all heart failure clinics will be able to contact the primary investigators with questions regarding the conduct of the trial. Heart failure clinics switch treatment strategies yearly. The heart failure clinics will be contacted 3-4 weeks prior to the scheduled annual switch-over to remind them of the upcoming switch-over. In addition, all heart failure clinics will receive stickers to put on the computer monitors, which state which strategy to use in the current period and when the next crossover occurs. To handle questions, all departments are offered a physical or online meeting before the annual switch-over.

Data collection during the allocation period No study-related data on individual patients will be collected during the allocation period, so there will be no case report forms.

Follow-up Patients will be followed according to the usual standard of care at their respective heart failure clinics. As there is no deviation from usual clinical practice except when to initiate MRA, patients will not be seen or followed as part of a study protocol. The treating physicians will discontinue treatment at their discretion according to usual practice. Discontinuation or cross-over will not exempt patients from the study, bring about additional procedures, and will not be reported to the sponsor-investigator. Hence, there will be no protocol-specific follow-up. Should new information emerge about one of the GDMTs, including information that changes the risk-benefit-ratio for patients or patient subgroups treated for heart failure, the patients will be informed about this via their local heart failure clinic.

For study-specific follow-up, data from the Danish Heart Failure Registry, which is routinely uploaded to Statistics Denmark, will be linked in anonymous form to hospital admissions, diagnoses, vital status, cause of death, dispensed descriptions, and biochemistry from The Danish National Patient Registry, The Danish Civil Registration System, The Clinical Laboratory Information System, and the Danish National Prescription Registry.

All patients will be followed up regardless of whether they adhere to the allocation arm, cross over to the other arm, or discontinue medication. Only patients who opt-out of the analysis will not be included in the follow-up.

Concomitant treatment No other treatments before, during, or after the trial will exempt patients from participation. Patients can be included in other research studies concomitantly and independently of this protocol.

Data management plan Data will be collected and processed in compliance with Regulation (EC) No 45/2001 and national data protection legislation implementing Regulation (EU) 2016/679, respectively. The trial is registered with the Knowledge Centre on Data Protection Compliance in Central Denmark Region. All data will be stored and analyzed on the Statistics Denmark servers through our agreement with the Division of Research Services at Statistics Denmark. Registration of patients who opt out of the study will be collected on paper and entered in a REDcap database. After the allocation period, before any analyses are performed, the REDcap database of patients who have opted out will be uploaded to the Statistics Denmark server and pseudo-anonymized. This will allow investigators to exclude patients who have opted out from all analyses. Data will be stored for 25 years after which opt out forms will be destroyed.

Source data All data will be collected from central Danish registries. Hence, there will be no case report forms; the only source data will be the opt-out forms from the patients who have opted out.

Analysis Primary endpoint The primary endpoint will be a combined endpoint of all-cause mortality or first hospitalization for worsening heart failure.

Secondary endpoints All-cause mortality First hospitalizations for heart failure Total hospitalizations Dialysis

Primary analysis Proportional hazard regression of time to the primary endpoint from the time of first claiming a prescription for HF medication, comparing strategy clusters adjusted for the department of cardiology.

Secondary analyses Cost-effectiveness analysis of each strategy. The proportion of patients who remained on MRA treatment for a minimum of one year.

Change in estimated glomerular filtration rate at one year. Difference in GDMT adherence Difference in patient reported outcome.

Patient cohort for analysis The patient cohort will consist of all patients registered in the Danish Heart Failure Registry during the allocation period with LVEF ≤40%, excluding patients who had opted out of the study.

Sample size considerations Based on data from the Danish Heart Failure Registry, investigators expect that approximately 4.000 patients will be enrolled in the heart failure registry annually. In the Danish Heart Failure Registry, 1-year mortality is ≈10%. With 24 clusters, four allocation periods and a mean cluster size per allocation period of 100 and assuming that 12% of patients in the control arm experience the primary outcome with an intraclass correlation of 0.03 and a cluster autocorrelation 0f 0.8, there will be a 91% power to detect a 15% reduction in the primary outcome in the intervention group.

Statistics Analyses will be performed according to the recommendation of the CONSORT statement for cluster trials. Primary results will be assessed as intention-to-treat. An instrumental variable analysis will be performed, where cluster randomization is used as an instrument for receiving treatment.

Results for subgroups will be presented. These will be prespecified before trial termination. Already planned subgroup analyses are age, gender, NYHA class, previous myocardial infarction, previous revascularization, hypertension, type 2 diabetes, chronic kidney disease stages, atrial fibrillation/flutter, and socio-economic status. A detailed statistical analysis plan will be prepared before study-termination.

Safety Patients will be treated according to standard clinical practice. Hence, the safety of the study participants is equal to that of patients who are not participating in the study.

All Danish heart failure clinics have strong experience initiating GDMT for HFrEF, including monitoring patient safety as part of common practice. Patients discharged from the outpatient clinics will be followed by their general practitioner with regular safety assessments as part of common practice. As patients are prescribed the same medical therapy, investigators do not expect any changes in the overall number of complications.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥18 years old who are newly diagnosed with HFrEF and allocated to an outpatient clinic for up-titration of guideline-directed medical therapy for HFrEF at participating cardiology departments

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16000 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Combined one year all-cause mortality or first hospitalization for worsening heart failure. | From date of enrollment until the date of first hospitalization for worsening heart failure or date of death from any cause, whichever comes first, assessed up to 200 months

SECONDARY OUTCOMES:
All-cause mortality | From date of enrollment until the date of first hospitalization for worsening heart failure or date of death from any cause, whichever comes first, assessed up to 200 months
First hospitalization for heart failure | From date of enrollment until the date of first hospitalization for worsening heart failure or date of death from any cause, whichever comes first, assessed up to 200 months
Total number of acute hospitalizations | From date of enrollment until the date of first hospitalization for worsening heart failure or date of death from any cause, whichever comes first, assessed up to 200 months
Need for dialysis | From date of enrollment until the date of first hospitalization for worsening heart failure or date of death from any cause, whichever comes first, assessed up to 200 months
Change in income | From date of enrollment until the date of first hospitalization for worsening heart failure or date of death from any cause, whichever comes first, assessed up to 200 months
  Change in income relative to pre-HFrEF, could be a surrogate marker of quality of life

IPD SHARING:
Plan to Share IPD: No
Study-participants will be followed using national Danish registers, and Danish legislation does not freely sharing of individual patient data